CLINICAL TRIAL: NCT02557386
Title: Optimal Volume of Bupivacaine in Adductor Canal Nerve Block in Patients Undergoing Unilateral Cruciate Ligament Reconstruction Surgery
Brief Title: Optimal Volume of Bupivacaine in Adductor Canal Nerve Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-001
Record Dates: First submitted 2015-09-11; First posted 2015-09-23 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia, Local
Keywords: Cruciate ligament surgery; Adductor canal; Nerve block
MeSH Terms: interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A Levobupivacaine 5 mL (Experimental): Adductor canal nerve block with levobupivacaine 0.25% 5 mL and perineural catheter placement, an elastomeric pump with bupivacaine 0.1% at a rate of 5 ml/hr will be placed after surgery for continuous nerve block.
  Interventions: Drug: Levobupivacaine 5 mL
- B Levobupivacaine 10 mL (Experimental): Adductor canal nerve block with levobupivacaine 0.25% 10 mL and perineural catheter placement, an elastomeric pump with bupivacaine 0.1% at a rate of 5 ml/hr will be placed after surgery for continuous nerve block.
  Interventions: Drug: Levobupivacaine 10 mL
- C Levobupivacaine 15 mL (Experimental): Adductor canal nerve block with levobupivacaine 0.25% 15 mL and perineural catheter placement, an elastomeric pump with bupivacaine 0.1% at a rate of 5 ml/hr will be placed after surgery for continuous nerve block.
  Interventions: Drug: Levobupivacaine 15 mL
- D Levobupivacaine 20 mL (Experimental): Adductor canal nerve block with levobupivacaine 0.25% 20 mL and perineural catheter placement, an elastomeric pump with bupivacaine 0.1% at a rate of 5 ml/hr will be placed after surgery for continuous nerve block.
  Interventions: Drug: Levobupivacaine 20 mL
- E Levobupivacaine 25 mL (Experimental): Adductor canal nerve block with levobupivacaine 0.25% 25 mL and perineural catheter placement, an elastomeric pump with bupivacaine 0.1% at a rate of 5 ml/hr will be placed after surgery for continuous nerve block.
  Interventions: Drug: Levobupivacaine 25 mL
- F Levobupivacaine 30 mL (Experimental): Adductor canal nerve block with levobupivacaine 0.25% 30 mL and perineural catheter placement, an elastomeric pump with bupivacaine 0.1% at a rate of 5 ml/hr will be placed after surgery for continuous nerve block.
  Interventions: Drug: Levobupivacaine 30 mL

INTERVENTIONS:
Drug: Levobupivacaine 5 mL — Levobupivacaine 0.25% 5 mL in adductor canal nerve block
  Other Names: Chirocaine
  Arms: A Levobupivacaine 5 mL
Drug: Levobupivacaine 10 mL — Levobupivacaine 0.25% 10 mL in adductor canal nerve block
  Other Names: Chirocaine
  Arms: B Levobupivacaine 10 mL
Drug: Levobupivacaine 15 mL — Levobupivacaine 0.25% 15 mL in adductor canal nerve block
  Other Names: Chirocaine
  Arms: C Levobupivacaine 15 mL
Drug: Levobupivacaine 20 mL — Levobupivacaine 0.25% 20 mL in adductor canal nerve block
  Other Names: Chirocaine
  Arms: D Levobupivacaine 20 mL
Drug: Levobupivacaine 25 mL — Levobupivacaine 0.25% 25 mL in adductor canal nerve block
  Other Names: Chirocaine
  Arms: E Levobupivacaine 25 mL
Drug: Levobupivacaine 30 mL — Levobupivacaine 0.25% 30 mL in adductor canal nerve block
  Other Names: Chirocaine
  Arms: F Levobupivacaine 30 mL

SUMMARY:
To establish adequate volume of levobupivacaine 0.25% in adductor canal nerve block in unilateral cruciate ligament of the knee reconstruction surgery.

DETAILED DESCRIPTION:
The complex knee surgery has been associated with severe postoperative pain. Different analgesic techniques for postoperative management of this increasingly common surgery, with main purpose of adequately control pain, minimizing adverse effects and seeking early rehabilitation.

Currently, the most used technique is the continuous femoral nerve block, which is able to control postoperative pain well, but has the limitation that also produces motor blockade, decreasing quadriceps strength up to 80%, increasing the number of falls and delaying early mobilization after surgery. On the other hand, the adductor canal nerve block is an alternative as it is considered a purely sensitive block. The nerves that are in this channel are the saphenous adductor nerve, posterior branches of the obturator nerve, medial vast nerve, sometimes the medial cutaneous nerve and anterior branches of the obturator nerve and the vast medial nerve.

With regard to the adductor canal block, current literature supports analgesic effect comparable to femoral nerve block with less motor block than femoral nerve block. However, there is no clarity regarding the ideal concentration and volume of local anesthetics to use. Volumes ranging from 5 to 30 ml have been used in different studies. For example, using 20 mL of local anesthetic in femoral nerve block has produced scattering of anesthetic that has blocked motor branches.

The investigators objective is to determine which volume of levobupivacaine 0.25% is necessary to produce analgesia and sensitive blockade while minimizing motor blockade in adductor canal nerve block in patients undergoing cruciate ligament reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* ASA status I or II
* BMI between 20 and 34 kg/m2
* Cruciate ligament of the knee reconstructive surgery
* No contraindications to general and regional anesthesia

Exclusion Criteria:

* Chronic pain more than 3 months
* Drug abuse
* Chronic use of analgesic drugs (more than 3 months)
* Psychiatric illness
* Peripheral neuropathy
* Drug allergy
* Severe gastroesophageal reflux disease

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in quadriceps motor force measured in kg*m/sec2 | Before nerve block (basal) and 24 hours after surgery
  Using a dynamometer in anterior tibial muscle

SECONDARY OUTCOMES:
Pain | Before surgery, 30 minutes after nerve block, one hour after surgery, 48 hours after surgery
  Using visual analogue scale, static and dynamic evaluation, scale from 0 (no pain) to 10 (worst pain imaginable)
Rescue analgesia | 24 hours and 48 hours after surgery
  Lidocaine 1% bolus through nerve block catheter and opioid use, measured in mg
Patient satisfaction | 48 hours after surgery
  Using a 5 point scale from 1 (very unsatisfied) to 5 (very satisfied)
Change in quadriceps force measured by 30-second chair stand test | Before nerve block (basal) and 24 hours after surgery
  Using 30-second chair stand test, how many times patient can stand up in 30 seconds, number of times is recorded
Sensitivity block | 30 minutes after adductor canal block
  Using a sensitivity scale ranging from 0 (no sensitivity), 1 (paresthesias) and 2 (normal sensitivity. Measured with needle prick and cold sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando R Altermatt, MD, Principal Investigator — Associate Professor Ordinary Category
Locations (1):
- Division de Anestesia - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Williams BA, Kentor ML, Vogt MT, Williams JP, Chelly JE, Valalik S, Harner CD, Fu FH. Femoral-sciatic nerve blocks for complex outpatient knee surgery are associated with less postoperative pain before same-day discharge: a review of 1,200 consecutive cases from the period 1996-1999. Anesthesiology. 2003 May;98(5):1206-13. doi: 10.1097/00000542-200305000-00024. PMID 12717143
- [Background] Grevstad U, Mathiesen O, Lind T, Dahl JB. Effect of adductor canal block on pain in patients with severe pain after total knee arthroplasty: a randomized study with individual patient analysis. Br J Anaesth. 2014 May;112(5):912-9. doi: 10.1093/bja/aet441. Epub 2014 Jan 8. PMID 24401802
- [Background] Capdevila X, Barthelet Y, Biboulet P, Ryckwaert Y, Rubenovitch J, d'Athis F. Effects of perioperative analgesic technique on the surgical outcome and duration of rehabilitation after major knee surgery. Anesthesiology. 1999 Jul;91(1):8-15. doi: 10.1097/00000542-199907000-00006. PMID 10422923
- [Background] Kim DH, Lin Y, Goytizolo EA, Kahn RL, Maalouf DB, Manohar A, Patt ML, Goon AK, Lee YY, Ma Y, Yadeau JT. Adductor canal block versus femoral nerve block for total knee arthroplasty: a prospective, randomized, controlled trial. Anesthesiology. 2014 Mar;120(3):540-50. doi: 10.1097/ALN.0000000000000119. PMID 24401769
- [Background] Allen HW, Liu SS, Ware PD, Nairn CS, Owens BD. Peripheral nerve blocks improve analgesia after total knee replacement surgery. Anesth Analg. 1998 Jul;87(1):93-7. doi: 10.1097/00000539-199807000-00020. PMID 9661553
- [Background] Hadzic A, Houle TT, Capdevila X, Ilfeld BM. Femoral nerve block for analgesia in patients having knee arthroplasty. Anesthesiology. 2010 Nov;113(5):1014-5. doi: 10.1097/ALN.0b013e3181f4b43d. No abstract available. PMID 20881593
- [Background] Charous MT, Madison SJ, Suresh PJ, Sandhu NS, Loland VJ, Mariano ER, Donohue MC, Dutton PH, Ferguson EJ, Ilfeld BM. Continuous femoral nerve blocks: varying local anesthetic delivery method (bolus versus basal) to minimize quadriceps motor block while maintaining sensory block. Anesthesiology. 2011 Oct;115(4):774-81. doi: 10.1097/ALN.0b013e3182124dc6. PMID 21394001
- [Background] Kandasami M, Kinninmonth AW, Sarungi M, Baines J, Scott NB. Femoral nerve block for total knee replacement - a word of caution. Knee. 2009 Mar;16(2):98-100. doi: 10.1016/j.knee.2008.10.007. Epub 2008 Nov 28. PMID 19046884
- [Background] Ilfeld BM, Duke KB, Donohue MC. The association between lower extremity continuous peripheral nerve blocks and patient falls after knee and hip arthroplasty. Anesth Analg. 2010 Dec;111(6):1552-4. doi: 10.1213/ANE.0b013e3181fb9507. Epub 2010 Oct 1. PMID 20889937
- [Background] Muraskin SI, Conrad B, Zheng N, Morey TE, Enneking FK. Falls associated with lower-extremity-nerve blocks: a pilot investigation of mechanisms. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):67-72. doi: 10.1016/j.rapm.2006.08.013. PMID 17196495
- [Background] Jaeger P, Grevstad U, Henningsen MH, Gottschau B, Mathiesen O, Dahl JB. Effect of adductor-canal-blockade on established, severe post-operative pain after total knee arthroplasty: a randomised study. Acta Anaesthesiol Scand. 2012 Sep;56(8):1013-9. doi: 10.1111/j.1399-6576.2012.02737.x. Epub 2012 Jul 26. PMID 22834681
- [Background] Krombach J, Gray AT. Sonography for saphenous nerve block near the adductor canal. Reg Anesth Pain Med. 2007 Jul-Aug;32(4):369-70. doi: 10.1016/j.rapm.2007.04.006. No abstract available. PMID 17720129
- [Background] Horn JL, Pitsch T, Salinas F, Benninger B. Anatomic basis to the ultrasound-guided approach for saphenous nerve blockade. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):486-9. doi: 10.1097/AAP.0b013e3181ae11af. PMID 19920424
- [Background] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014
- [Background] Lund J, Jenstrup MT, Jaeger P, Sorensen AM, Dahl JB. Continuous adductor-canal-blockade for adjuvant post-operative analgesia after major knee surgery: preliminary results. Acta Anaesthesiol Scand. 2011 Jan;55(1):14-9. doi: 10.1111/j.1399-6576.2010.02333.x. Epub 2010 Oct 29. PMID 21039357
- [Background] Jaeger P, Nielsen ZJ, Henningsen MH, Hilsted KL, Mathiesen O, Dahl JB. Adductor canal block versus femoral nerve block and quadriceps strength: a randomized, double-blind, placebo-controlled, crossover study in healthy volunteers. Anesthesiology. 2013 Feb;118(2):409-15. doi: 10.1097/ALN.0b013e318279fa0b. PMID 23241723
- [Background] Kwofie MK, Shastri UD, Gadsden JC, Sinha SK, Abrams JH, Xu D, Salviz EA. The effects of ultrasound-guided adductor canal block versus femoral nerve block on quadriceps strength and fall risk: a blinded, randomized trial of volunteers. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):321-5. doi: 10.1097/AAP.0b013e318295df80. PMID 23788068
- [Background] Saranteas T, Anagnostis G, Paraskeuopoulos T, Koulalis D, Kokkalis Z, Nakou M, Anagnostopoulou S, Kostopanagiotou G. Anatomy and clinical implications of the ultrasound-guided subsartorial saphenous nerve block. Reg Anesth Pain Med. 2011 Jul-Aug;36(4):399-402. doi: 10.1097/AAP.0b013e318220f172. PMID 21697687
- [Background] Chen J, Lesser JB, Hadzic A, Reiss W, Resta-Flarer F. Adductor canal block can result in motor block of the quadriceps muscle. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):170-1. doi: 10.1097/AAP.0000000000000053. PMID 24553306
- [Background] Davis JJ, Bond TS, Swenson JD. Adductor canal block: more than just the saphenous nerve? Reg Anesth Pain Med. 2009 Nov-Dec;34(6):618-9. doi: 10.1097/AAP.0b013e3181bfbf00. No abstract available. PMID 19901788
- [Background] Choi S, Trang A, McCartney CJ. Reporting functional outcome after knee arthroplasty and regional anesthesia: a methodological primer. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):340-9. doi: 10.1097/AAP.0b013e318295d973. PMID 23788070
- [Background] Bohannon RW. Measuring knee extensor muscle strength. Am J Phys Med Rehabil. 2001 Jan;80(1):13-8. doi: 10.1097/00002060-200101000-00004. PMID 11138949
- [Background] Jaeger P, Koscielniak-Nielsen ZJ, Schroder HM, Mathiesen O, Henningsen MH, Lund J, Jenstrup MT, Dahl JB. Adductor canal block for postoperative pain treatment after revision knee arthroplasty: a blinded, randomized, placebo-controlled study. PLoS One. 2014 Nov 11;9(11):e111951. doi: 10.1371/journal.pone.0111951. eCollection 2014. PMID 25386752
- [Background] Munoz HR, Cortinez LI, Altermatt FR, Dagnino JA. Remifentanil requirements during sevoflurane administration to block somatic and cardiovascular responses to skin incision in children and adults. Anesthesiology. 2002 Nov;97(5):1142-5. doi: 10.1097/00000542-200211000-00018. PMID 12411799
- [Background] Bouvet L, Da-Col X, Chassard D, Dalery F, Ruynat L, Allaouchiche B, Dantony E, Boselli E. ED(5)(0) and ED(9)(5) of intrathecal levobupivacaine with opioids for Caesarean delivery. Br J Anaesth. 2011 Feb;106(2):215-20. doi: 10.1093/bja/aeq296. Epub 2010 Oct 30. PMID 21037268